CLINICAL TRIAL: NCT01900821
Title: National Mammography Database
Status: Recruiting | Type: Observational
Sponsor: American College of Radiology (Other)
Responsible Party: Sponsor
Other Study IDs: NRDR-NMD
Record Dates: First submitted 2013-07-11; First posted 2013-07-17 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Screening and Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women: All women having mammograms

SUMMARY:
The National Mammography Database (NMD) leverages data that radiology practices are already collecting under federal mandate by providing them with comparative information for national and regional benchmarking. Participants receive semi-annual feedback reports that include important benchmark data such as cancer detection rates, positive predictive value rates and recall rates. Participation in the NMD is free to Breast Imaging Center of Excellence (BICOE) facilities.

ELIGIBILITY:
Inclusion Criteria:

* All

Exclusion Criteria:

* None

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women (primarily, but not exclusively), having mammograms at facilities participating in the registry
Sampling Method: Non-Probability Sample
Enrollment: 8000000 (Estimated)
Dates: Start 2009-07; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cancer Detection Rate | 1 year
  This outcome measure is measured using one year of follow-up after a mammogram is performed on a woman, and is aggregated by interpreting physician. Because the NMD is a registry and screening mammograms are annual exams for most patients, this measure is calculated each year using one year of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- ACR, Reston, Virginia, United States